CLINICAL TRIAL: NCT02073136
Title: Effect of a Phosphate Modified Diet on Phosphate Balance and Phosphate Metabolism in Predialysis Patients Stage 3-4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Camilla Storm Slumstrup (Unknown); Ewa Lewin (Unknown); Casper Rydahl (Unknown)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate professor at the University of Copenhagen, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2013-106
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phosphate modified diet (Experimental)
  Interventions: Other: Diet with phosphate containing additives; Other: Diet without phosphate containing additives

INTERVENTIONS:
Other: Diet with phosphate containing additives
Other: Diet without phosphate containing additives

SUMMARY:
Patients with chronic kidney disease struggle to eliminate phosphate as the renal function deteriorates, which results in accumulation of phosphate in the body. This has been shown to increase the patients' risk of cardiovascular disease and death. Even with dialysis treatment the patients cannot excrete enough phosphate to reach phosphate balance. The patients are therefore recommended a very restrictive diet when they reach the dialysis stage. It is therefore important to find ways to prevent such accumulation of phosphate in the body as early in the disease process as possible, but without compromising the nutritional status. Because phosphate occurs naturally in many of our foods, such as meat, fish and dairy products, it is difficult to reduce the intake of phosphate, without also reducing the intake of energy and protein. Over the past couple of years there has been an increased focus on the use of phosphate containing additives in the food industry. A reduction in the intake of phosphorus containing additives may reduce the accumulation of phosphate in the body. This can be achieved by decreasing the intake of processed food products. Because it is also very time consuming and inconvenient for the patient to keep these strict diets, the patients have a reasonable claim to know which effects can be achieved by such diets. This will therefore seek to be further explored in the following study. The study is conducted as a randomised crossover trial in predialysis patients stage 3-4.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years.
* Diagnosed with Chronic Kidney Disease stage 3-4 (GFR 15-59 ml / min)
* p-phosphate between 0.85 mmol / L (2.7 mg / dL) and 1.50 mmol / L (4.7 mg / dl)
* Read and understand Danish
* Have received oral and written information about the study
* Signed informed consent form

Exclusion Criteria:

* Diagnosed hyperphosphatemia
* Diagnosed hyperparathyroidism
* Treatment with phosphate binders
* Dysphagia
* Diagnosed with decreased absorption capacity in the intestine
* Co-morbidities in liver, pancreas or lungs
* Dementia
* Pregnancy / breastfeeding
* Embedded within the last 4 weeks
* Kidney transplant
* Terminal patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Phosphate balance | 1 week

SECONDARY OUTCOMES:
p-phosphate | 1 week
p-PTH | 1 week
p-Calcium | 1 week
FGF23 | 1 week
p-25(OH)D | 1 week
Calcium-phosphate product | 1 week
p-alkaline phosphatase | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD, MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Herlev Hospital, Herlev, Herlev Ringvej 75, Denmark